CLINICAL TRIAL: NCT04528043
Title: Infections and Colonization With the Third Group of Enterobacteriaceae in the Intensive Care Impact on the Mortality and Morbidity
Brief Title: Infections and Colonization With the Third Group of Enterobacteriaceae in the Intensive Care Unit
Acronym: EB3REA
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: PSS2018/EB3REA-NOVY/YB
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-02

CONDITIONS: Critically Ill; Enterobacteriaceae Infections; Antibiotic Resistant Infection
Keywords: Third group Enterobacteriaceae; infection; colonization; resistance; AMPc cephalosporinase
MeSH Terms: conditions — Critical Illness; Enterobacteriaceae Infections; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- critically ill patients: critically ill patients admitted in one of the 5 ICUs of the university hospital of Nancy during the year 2016 with documented third group enterobacteriaceae infection and/or colonization with third group enterobacteriaceae

SUMMARY:
There is a lack of data whether colonization and infection with Enterobacteriaceae of the third group (EB3) affect the outcomes for ICU patients. This study evaluated the effects of EB3 colonization and infection on ICU mortality, ICU length of stay (LOS) and broad-spectrum antibiotic exposure. We focused on the sub type Enterobacter regarding its a priori higher risk of resistance.

ELIGIBILITY:
Inclusion Criteria:

* adults critically ill patients admitted to the the participating ICUs during the study period
* with colonization and/or infection with a third group enterobacteriacea
* and with a lenght of stay > 24h

Exclusion Criteria:

* minors patients
* lenght of stay < 24h

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults (≥ 18 years-old) patients admitted in the participating ICUs with LOS ≥ 24 hours during the study period were enrolled if they had presented a colonization and/or an infection caused by an EB3 (Enterobacter cloacae, Enterobacter aerogenes, Morganella morganii, Serratia marcescens, Hafnia alvei et Citrobacter freundii), from 1st January 2016 to 31th December 2016.
  Participating ICUs of the university hospital of Nancy:
  * two Medical ICU
  * 3 surgical ICU
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
all cause mortality | Day 180
  Evaluation of the impact of colonization and/or infection with third group enterobacteriaceae on mortality during hospitalization and up to 180 day

SECONDARY OUTCOMES:
Resistance strains of sub type enterobacter | DAY 90
  Evaluation of number of resistant strains among Enterobacter subtype in comparison with other third group enterobacteriaceae

CONTACTS AND LOCATIONS:
Locations (1):
- Emmanuel NOVY, Vandœuvre-lès-Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: No